CLINICAL TRIAL: NCT03987477
Title: Brief Online Intervention to Modify Interpretation Biases in Depression: An Experimental Approach
Brief Title: Online Intervention to Modify Interpretation Biases in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT17/17-CT18/17 UCM
Record Dates: First submitted 2019-06-07; First posted 2019-06-17 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Depression; Cognitive Change
Keywords: Cognitive Biases; Cognitive Bias Modification; Depression; Online intervention; Cognitive Bias Interpretation
MeSH Terms: conditions — Depression | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will be exposed to a brief online program aimed at the modification of negative emotional cognitive biases. The program consists of an introduction and four 1-hour sessions, in video format. In each session, participants are required to complete some open questions and scales about the type of cognitive bias addressed in each session. All sessions are structured in four parts: 1) description and examples of some specific cognitive biases; 2) information about negative consequences of each bias; 3) explanation of adaptive strategies to modify cognitive biases (i.e., the four-questions approach used in standard Cognitive behavioral therapy); and 4) use of some practices to familiarize participants with the use of those strategies.
  Interventions: Behavioral: Interpretation bias modification program
- Waiting list group (Other): The control group will be composed of individuals waiting for the treatment. Participants will not be exposed to the experimental program or any other between the pre-evaluation and the post-evaluation sessions. Participants in this group will have access to the potential benefits of the intervention after the post-evaluation of both groups.
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: Interpretation bias modification program — Brief online program aimed at the modification of negative interpretation biases.
  Other Names: Cognitive bias modification; Online cognitive bias intervention; Online interpretation bias intervention
  Arms: Experimental group
Behavioral: Waiting list — Waiting list procedure for the control group.
  Arms: Waiting list group

SUMMARY:
Cognitive biases have been found to be possible causal and vulnerability factors for depression. There is empirical evidence on the presence of negative emotional biases in interpretation in people with depressive symptoms. A whole new area of research, called Cognitive Bias Modification (CBM), is focused on targeting negative cognitive emotional biases to investigate its impact on clinical symptoms. A recent meta-analysis has shown that this type of programs are effective in reducing cognitive biases but there is still controversy on their clinical value to reduce symptoms. The purpose of the study is to create a brief online intervention aimed to reduce negative emotional cognitive biases present in depression and to analyze its impact on clinical symptoms and well-being.

DETAILED DESCRIPTION:
More specifically, the intervention is framed within the area of CBM but it is rooted on techniques and change procedures used in cognitive-behavioral therapies. While original CBM studies train participants to change cognitive biases in an automatic manner, by forcing individuals to find positive outcomes to ambiguous scenarios, this new intervention focuses on teaching participants the meaning of emotional cognitive biases and how to modify them by using an effortful type of processing (i.e., looking for adaptive alternative interpretations to ambiguous stories).

The study has been design to overcome some of the limitations that have been pointed out in this emerging research area. Firstly, although there are recent efforts to understand how interpretation, attention and memory cognitive biases may be related, it is still not clear how they interact with each other. For this purpose, some authors have pointed out the need to use longitudinal data to see how one process may affect each other over time. Secondly, different systematic reviews and meta-analyses have investigated the moderating role of variables that may be affecting the heterogeneity of results found in CBM interventions. Mental imagery has been found to be a useful tool to help participants in their changing process, while there is no preferred number of sessions for these interventions. This study will help shed some light into this factors by using mental imagery during four sessions online.

ELIGIBILITY:
Inclusion Criteria:

* Present (PHQ-9) or past (DID) episode of depression.
* Access to Internet
* Fluent in Spanish language

Exclusion Criteria:

* Being under any psychological treatment
* Having a psychotic condition
* Having any cognitive impairment or condition that do not allow to follow the program
* Serious auditory or visual impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Total score of pleasantness ratings given to the ambiguous scenarios presented in the Ambiguous Scenarios Test for Depression-II, (AST-D-II) to measure interpretation bias. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention) and the follow-up assessments (2 weeks and 3 months after completing the intervention).
  Participants are asked to rate how pleasant they perceive 15 ambiguous scenarios in a scale from -5 (very unpleasant) to 5 (very pleasant).
Total score of each of the three subscales of the Depression, Anxiety and Stress Scale-21 (DASS) questionnaire. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention) and the follow-up assessments (2 weeks and 3 months after completing the intervention).
  Three subscales, with 7 items each, measuring symptoms of depression, anxiety and stress. Scores multiplied by 2 and summed up for each scale.
Total score on general, eudaimonic, hedonic, and social well-being as measured by the Pemberton Happiness Index (PHI) | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention) and the follow-up assessments (2 weeks and 3 months after completing the intervention).
  Scale of 11 items measuring emotional well-being at different levels.

SECONDARY OUTCOMES:
Ratio of the number of negative unscrambled sentences by the number of emotional unscrambled sentences in the Scrambled Sentence Test (SST) with cognitive load. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  The task presents 20 scrambled sentences with 6 words each. Participants are asked to construct a sentence using 5 of the 6 words. In addition, participants are shown a number, at the beginning of the task, to report it at the end (cognitive load). The resulting ratio of correctly negative unscrambled sentences between correctly emotional unscrambled sentences is an index of automatic interpretation bias.
Proportion of time fixating the mouse cursor on negative over positive words to uncover them during the SST. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  During the SST, words are covered so that participants can only see them when placing the mouse cursor over them. The time spent on negative words is a measure of negative attention bias.
Ratio of recalled negative unscrambled sentences and recalled emotional unscrambled sentences during the SST. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  Participants are asked to remember, during 5 minutes, the sentences they construct during the SST. The ratio of negative and emotional unscrambled sentences that participants recall is a measure of memory bias.
Number of items viewed before reaching a decision in the Computerized Beads Task. | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  The task presents two jars with beads containing positive or negative adjectives. Each jar has a different ratio of positive and negative words. Participants are told that one of the jars is going to be selected and one bead is going to be taken out and returned to it in each trial. Participants have to decide which jar is being used based on the number of positive and negative adjectives that are taken in each trial. The number of beads viewed before reaching a decision is an index of jumping to conclusion bias.
Total score on the Dysfunctional Attitudes Scale (DAS) | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  Scale of 40 sentences which participants have to rate from 1 (totally agree) to 7 (totally disagree). The sum of the scores given to each sentence is an index of dysfunctional cognitive schemas.
Total score on the Brooding subscale of the Ruminative Responses Scale (RRS) | Change from the first assesment (the day before starting the intervention) to the second assessment (the day after completing the intervention).
  Subscale of 5 items which participants have to rate from 1 (totally disagree) to 5 (totally agree). The total score, ranging from 5 to 25, is an index of brooding.

OTHER OUTCOMES:
Four of more depressive symptoms (including anhedonia and depressed modd) in the Patient Health Questionnaire-9 (PHQ-9) | Screening measure used after potential participants contact the main researcher to collaborate and before selecting participants to include in the study.
  9 items measuring symptoms of depression from 1 (not at all) to 4 (nearly everyday). Diagnosis is made if participants select 3 o 4 in four or more items (including anhedonia and depressed mood).
Five of more depressive symptoms (including anhedonia and depressed modd) in the Diagnostic Inventory of Depression (DID). | Screening measure used after potential participants contact the main researcher to collaborate and before selecting participants to include in the study.
  Scale of 42 items measuring symptoms of depression in the past from 0 to 4.
Total score in each of the 5 subscales of the EVEA assessment of current mood. | Participants self-administer the scale right before each session at home and right after completing each session.
  Participants have to rate, from 0 to 10, their current level of anger, happiness, anxiety, depression, and boredom. Scores of each subscale (4 items each) are summed up.
Total number of events, total number of times, mean score on negative impact and mean duration time of the negative impact of the negative events selected in the Stressful events questionnaire (based on Life Events Scale, LES). | The questionnaire is used 2 weeks and 3 moths after finishing the program (follow-ups).
  A 47-item questionnaire in which participants select negative events they have experienced during the last two weeks or three months, the number of times each event was experienced, the emotional impact of the event and the duration time of the emotional impact. The different indexes represent experience of stressful events.
Total score on each of the two subscales (treatment expectancy and rationale credibility) of the Credibility and expectancy questionnaire (CEQ) | This scale is administered the day before starting the intervention.
  6 items measuring patients' expectancy of treatment success and credibility of the treatment prior to the intervention.
Total score on the Client Satisfaction Questionnaire (CSQ-8) | The measure is administered one day after finishing the intervention.
  8 items measuring participants' satisfaction with the treatment rated with a 4-point scale where 1 reflects 'very low satisfaction' and 4 reflects 'very high satisfaction'.

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Vázquez, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Faculty of Psychology, Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The authors have not decided yet on IPD sharing.

REFERENCES:
- [Background] Becker, E. S., & Vrijsen, J. N. Cognitive processes in CBT. In The science of cognitive behavioral therapy (pp. 77-106). Academic Press, 2017
- [Background] Everaert J, Koster EH, Derakshan N. The combined cognitive bias hypothesis in depression. Clin Psychol Rev. 2012 Jul;32(5):413-24. doi: 10.1016/j.cpr.2012.04.003. Epub 2012 Apr 21. PMID 22681914
- [Background] Gotlib IH, Joormann J. Cognition and depression: current status and future directions. Annu Rev Clin Psychol. 2010;6:285-312. doi: 10.1146/annurev.clinpsy.121208.131305. PMID 20192795
- [Background] Jones EB, Sharpe L. Cognitive bias modification: A review of meta-analyses. J Affect Disord. 2017 Dec 1;223:175-183. doi: 10.1016/j.jad.2017.07.034. Epub 2017 Jul 18. PMID 28759865
- [Background] Sanchez, A., Duque, A., Romero, N., & Vazquez, C. Disentangling the interplay among cognitive biases: Evidence of combined effects of attention, interpretation and autobiographical memory in depression. Cognitive Therapy and Research 41(6): 829-841, 2017.
- [Background] Everaert J, Duyck W, Koster EH. Attention, interpretation, and memory biases in subclinical depression: a proof-of-principle test of the combined cognitive biases hypothesis. Emotion. 2014 Apr;14(2):331-40. doi: 10.1037/a0035250. Epub 2014 Feb 10. PMID 24512247
- [Background] Duque, A., López-Gómez, I., Blanco, I., & Vázquez, C. Modificación de Sesgos Cognitivos (MSC) en depresión: Una revisión crítica de nuevos procedimientos para el cambio de sesgos cognitivos. Terapia Psicológica 33(2): 103-116, 2015
- [Background] Menne-Lothmann C, Viechtbauer W, Hohn P, Kasanova Z, Haller SP, Drukker M, van Os J, Wichers M, Lau JY. How to boost positive interpretations? A meta-analysis of the effectiveness of cognitive bias modification for interpretation. PLoS One. 2014 Jun 26;9(6):e100925. doi: 10.1371/journal.pone.0100925. eCollection 2014. PMID 24968234
- [Background] Cristea IA, Kok RN, Cuijpers P. Efficacy of cognitive bias modification interventions in anxiety and depression: meta-analysis. Br J Psychiatry. 2015 Jan;206(1):7-16. doi: 10.1192/bjp.bp.114.146761. PMID 25561486
- [Derived] Nieto I, Vazquez C. Disentangling the mediating role of modifying interpretation bias on emotional distress using a novel cognitive bias modification program. J Anxiety Disord. 2021 Oct;83:102459. doi: 10.1016/j.janxdis.2021.102459. Epub 2021 Jul 29. PMID 34358756
- [Derived] Nieto I, Vazquez C. 'Relearning how to think': A brief online intervention to modify biased interpretations in emotional disorders-study protocol for a randomised controlled trial. Trials. 2021 Jul 31;22(1):510. doi: 10.1186/s13063-021-05459-3. PMID 34332616